CLINICAL TRIAL: NCT01018888
Title: Clinical Assessment of Auro KPro
Brief Title: Safety and Efficacy Study of Artificial Cornea
Acronym: AuroKPro
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1010941
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2011-07

CONDITIONS: Corneal Transplantation
Keywords: Cornea; Transplantation, Cornea; Keratoplasty; Grafting, Corneal
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Keratoprosthesis (Experimental)
  Interventions: Device: Auro KPro (Keratoprosthesis)

INTERVENTIONS:
Device: Auro KPro (Keratoprosthesis) — Front plate with optical cylinder, a back plate and a titanium ring to hold the complex together
  Other Names: Auro KPro

SUMMARY:
The purpose of this study is to evaluate the stability of artificial cornea manufactured by Aurolab and to assess its visual outcomes.

DETAILED DESCRIPTION:
The keratoprosthesis, also know as an artificial cornea plays a significant role in combating corneal blindness in patients who are no longer candidates for penetrating keratoplasty.The global incidence of corneal blindness is estimated to be 6-8 million. In India there are approximately 6.8 million cases of unilateral corneal blindness and 1.3 million people with bilateral corneal pathology.

Eligible subjects after getting informed consent will be included in this study. All the subjects will have pre-operative evaluation which includes history, visual acuity, Intraocular pressure (IOP), evaluation of tear film and ultrasound A and B scan. Ocular inflammation will be controlled prior to surgery. Keratoplasty will be performed with keratoprosthesis under local anesthesia. Patients will be followed up at regular interval to assess the outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years
* Willing to participate and review on schedule
* Multiple failed grafts with poor prognosis for regrafting
* Adequate tear film and lid function
* Projection of light in all quadrants
* Bilateral blind

Exclusion Criteria:

* Reasonable chance of success with keratoplasty
* Autoimmune disease such as Stevens Johnson Syndrome, Pemphigoid
* End stage glaucoma
* Retinal detachment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1st Month, 2nd Month, 3rd Month,5th Month, 7th Month, 9th Month and 12th Month

SECONDARY OUTCOMES:
Retention of the device | 1st Month, 2nd Month, 3rd Month,5th Month, 7th Month, 9th Month and 12th Month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jeena Mascarenhas, MBBS, MS, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India